CLINICAL TRIAL: NCT00106002
Title: A Phase II Study of Alimta as First Line Chemotherapy for Advanced or Metastatic Breast Cancer
Brief Title: Pemetrexed as the First Treatment in Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9028; H3E-US-S045
Record Dates: First submitted 2005-03-18; First posted 2005-03-21 (Estimated); Results first posted 2009-06-01 (Estimated); Last update posted 2009-06-01 (Estimated); Status verified 2009-04

CONDITIONS: Breast Cancer; Breast Neoplasms, Male; Carcinoma, Ductal
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male; Carcinoma, Ductal | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Drug: pemetrexed

INTERVENTIONS:
Drug: pemetrexed — 600 mg/m2, intravenous (IV), every 14 days until complete response or disease progression
  Other Names: LY231514; Alimta

SUMMARY:
The purposes of this study are to determine whether pemetrexed can help patients with metastatic (cancer that has spread to other parts of the body) breast cancer, to determine any side effects that may be associated with the drug, to determine how much pemetrexed should be given to patients, and to collect DNA for future research regarding metastatic breast cancer. The collection of DNA is optional to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Must have been diagnosed with either advanced or metastatic breast cancer.
* Chemotherapy has not been given for advanced or metastatic breast cancer.
* The diagnosis of advanced or metastatic breast cancer was made at least 12 months after chemotherapy was given after breast surgery.
* Able to carry out work of a light nature (for example, light housework, office work).
* Must be at least 18 years old.

Exclusion Criteria:

* Have received prior bone marrow or peripheral stem cell transplantation.
* Have received prior chemotherapy for metastatic breast cancer.
* Are currently pregnant or breast-feeding.
* Have an active infection that your doctor decides will affect your safety.
* Are unable to take folic acid or vitamin B12.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pemetrexed
Started | 37
Completed | 35 (Completed means that the patient was evaluable for response.)
Not Completed | 2
Not completed — Did not take any study drug | 1
Not completed — Ineligible after Registration | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed
Number analyzed (Participants) | 37
Age Continuous [Median (Full Range); unit: years] | 61.4 [39 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 37
Eastern Cooperative Oncology Group Scale Performance Status [Number; unit: participants]
  0 - Fully Active | 19
  1 - Ambulatory, Restricted Strenuous Activity | 18
  2 - Ambulatory, No Work Activities | 0
  3 - Partially Confined to Bed, Limited Self Care | 0
  4 - Completely Disabled | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Tumor Response
Description: Best response recorded from the start of treatment until disease progression/recurrence using Response Evaluation Criteria In Solid Tumors (RECIST) criteria that defines when participants improve ("respond"), stay the same ("stable"), or worsen ("progression") during treatment.
Time Frame: every 3 cycles (approximately 6-7 weeks) or until patient has disease progression
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 35
participants
  Complete Response | 1
  Partial Response | 8
  Stable Disease | 14
  Progressive Disease | 9
  Best Response Not Evaluable | 3

2. Secondary Outcome: Toxicity Profile: Adverse Events (Common Terminology Criteria for Adverse Events, Grade 3 and 4, Present in >5% of Participants)
Description: Participants rated for toxicity prior to each cycle using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events v3.0 (CTCAE). Grades range from 0 (no AE or within normal limits) to 5 (death related to AE).
Time Frame: every 14 day cycle, and during 30-days post-therapy follow-up and long-term follow-up
Measure: Number; unit: participants
Arm/Group | Pemetrexed
Number analyzed (Participants) | 36
participants
  Anaemia - Grade 3 | 5
  Anaemia - Grade 4 | 0
  Leukopenia - Grade 3 | 4
  Leukopenia - Grade 4 | 2
  Neutropenia - Grade 3 | 8
  Neutropenia - Grade 4 | 5
  Constipation - Grade 3 | 2
  Constipation - Grade 4 | 0
  Nausea - Grade 3 | 3
  Nausea - Grade 4 | 0
  Asthenia - Grade 3 | 3
  Asthenia - Grade 4 | 0
  Fatigue - Grade 3 | 5
  Fatigue - Grade 4 | 0
  Cellulitis - Grade 3 | 2
  Cellulitis - Grade 4 | 0
  Dehydration - Grade 3 | 2
  Dehydration - Grade 4 | 0
  Hyperglycaemia - Grade 3 | 3
  Hyperglycaemia - Grade 4 | 2
  Dyspnoea - Grade 3 | 4
  Dyspnoea - Grade 4 | 0
  Pleural effusion - Grade 3 | 2
  Pleural effusion - Grade 4 | 0

3. Secondary Outcome: Duration of Tumor Response
Description: Defined as time from first observation of complete response or partial response to the first observation of progressive disease or death due to any cause.
Time Frame: every 3 cycles (approximately 6-7 weeks) or until patient has disease progression
Population: Only applies to patients who had a complete or partial response
Measure: Median (Full Range); unit: months
Arm/Group | Pemetrexed
Number analyzed (Participants) | 9
months | 7.3 [3.0 to 20.6]

4. Secondary Outcome: Progression-Free Survival Time
Description: Defined as the time from date of first dose to the first observation of disease progression, or death due to any cause.
Time Frame: every 3 cycles (approximately 6-7 weeks) or until patient has disease progression
Population: Intent to treat population (in order to follow protocol, one patient who did not take study drug was excluded from this analysis)
Measure: Median (Full Range); unit: months
Arm/Group | Pemetrexed
Number analyzed (Participants) | 36
months | 4.1 [0.5 to 22.4]

5. Secondary Outcome: Overall Survival Time
Description: Defined as the time from date of first dose to time of death due to any cause.
Time Frame: every 14 day cycle, during 30-days post-therapy follow-up, and every 6 months during the long-term follow-up
Population: Intent to treat population (in order to follow protocol, one patient who did not take any study drug was excluded from this analysis)
Measure: Median (Full Range); unit: months
Arm/Group | Pemetrexed
Number analyzed (Participants) | 36
months | 18.9 [0.5 to 27.7]

ADVERSE EVENTS:
Groups:
- Pemetrexed: Pemetrexed
Arm/Group | Pemetrexed
Serious Adverse Events (participants affected / at risk) | 14
Other Adverse Events (participants affected / at risk) | 34
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Pemetrexed
Anaemia (Blood and lymphatic system disorders) | 2/36 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1/36 (1)
Angina pectoris (Cardiac disorders) | 1/36 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1/36 (1)
Diarrhoea (Gastrointestinal disorders) | 1/36 (1)
Nausea (Gastrointestinal disorders) | 3/36 (3)
Vomiting (Gastrointestinal disorders) | 2/36 (2)
Asthenia (General disorders) | 1/36 (1)
Fatigue (General disorders) | 1/36 (1)
Cellulitis (Infections and infestations) | 2/36 (5)
Peritonitis bacterial (Infections and infestations) | 1/36 (1)
Upper respiratory tract infection (Infections and infestations) | 1/36 (1)
Urinary tract infection (Infections and infestations) | 1/36 (1)
Blood creatinine increased (Investigations) | 1/36 (1)
Nutritional condition abnormal (Investigations) | 1/36 (1)
Dehydration (Metabolism and nutrition disorders) | 1/36 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1/36 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1/36 (1)
Dizziness (Nervous system disorders) | 2/36 (2)
Mental status changes (Psychiatric disorders) | 2/36 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1/36 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2/36 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2/36 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1/36 (1)
Lymphoedema (Vascular disorders) | 1/36 (2)
Visceral arterial ischaemia (Vascular disorders) | 1/36 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Pemetrexed
Anaemia (Blood and lymphatic system disorders) | 26/36 (78)
Leukopenia (Blood and lymphatic system disorders) | 12/36 (36)
Lymphopenia (Blood and lymphatic system disorders) | 3/36 (4)
Neutropenia (Blood and lymphatic system disorders) | 21/36 (51)
Thrombocytopenia (Blood and lymphatic system disorders) | 6/36 (10)
Palpitations (Cardiac disorders) | 2/36 (2)
Tachycardia (Cardiac disorders) | 3/36 (3)
Eye irritation (Eye disorders) | 2/36 (2)
Lacrimation increased (Eye disorders) | 2/36 (2)
Vision blurred (Eye disorders) | 3/36 (3)
Abdominal pain (Gastrointestinal disorders) | 7/36 (7)
Ascites (Gastrointestinal disorders) | 2/36 (2)
Constipation (Gastrointestinal disorders) | 10/36 (13)
Diarrhoea (Gastrointestinal disorders) | 9/36 (13)
Dry mouth (Gastrointestinal disorders) | 2/36 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2/36 (2)
Nausea (Gastrointestinal disorders) | 18/36 (41)
Oral pain (Gastrointestinal disorders) | 2/36 (2)
Stomatitis (Gastrointestinal disorders) | 2/36 (2)
Vomiting (Gastrointestinal disorders) | 9/36 (16)
Asthenia (General disorders) | 6/36 (11)
Chills (General disorders) | 2/36 (2)
Fatigue (General disorders) | 26/36 (47)
Generalised oedema (General disorders) | 3/36 (5)
Mucosal inflammation (General disorders) | 4/36 (5)
Oedema peripheral (General disorders) | 8/36 (12)
Pain (General disorders) | 2/36 (3)
Pyrexia (General disorders) | 5/36 (7)
Cellulitis (Infections and infestations) | 3/36 (5)
Rhinitis (Infections and infestations) | 2/36 (2)
Sinusitis (Infections and infestations) | 4/36 (5)
Upper respiratory tract infection (Infections and infestations) | 3/36 (3)
Urinary tract infection (Infections and infestations) | 5/36 (7)
Contusion (Injury, poisoning and procedural complications) | 3/36 (3)
Alanine aminotransferase (Investigations) | 2/36 (3)
Alanine aminotransferase increased (Investigations) | 10/36 (16)
Aspartate aminotransferase (Investigations) | 2/36 (3)
Aspartate aminotransferase increased (Investigations) | 9/36 (17)
Blood alkaline phosphatase increased (Investigations) | 4/36 (7)
Blood glucose increased (Investigations) | 2/36 (7)
Blood lactate dehydrogenase increased (Investigations) | 3/36 (3)
Weight decreased (Investigations) | 4/36 (5)
White blood cell count increased (Investigations) | 2/36 (3)
Anorexia (Metabolism and nutrition disorders) | 11/36 (16)
Decreased appetite (Metabolism and nutrition disorders) | 2/36 (2)
Dehydration (Metabolism and nutrition disorders) | 2/36 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 8/36 (21)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3/36 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 3/36 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 2/36 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3/36 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4/36 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2/36 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 5/36 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3/36 (4)
Coordination abnormal (Nervous system disorders) | 2/36 (2)
Dizziness (Nervous system disorders) | 7/36 (9)
Dysgeusia (Nervous system disorders) | 2/36 (2)
Headache (Nervous system disorders) | 8/36 (8)
Paraesthesia (Nervous system disorders) | 3/36 (4)
Tremor (Nervous system disorders) | 2/36 (2)
Anxiety (Psychiatric disorders) | 5/36 (5)
Depression (Psychiatric disorders) | 5/36 (7)
Insomnia (Psychiatric disorders) | 8/36 (8)
Breast pain (Reproductive system and breast disorders) | 2/36 (2)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2/36 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5/36 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9/36 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2/36 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2/36 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 4/36 (4)
Erythema (Skin and subcutaneous tissue disorders) | 3/36 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2/36 (2)
Rash (Skin and subcutaneous tissue disorders) | 10/36 (13)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2/36 (2)
Swelling face (Skin and subcutaneous tissue disorders) | 2/36 (2)
Hot flush (Vascular disorders) | 4/36 (4)
Hypotension (Vascular disorders) | 2/36 (2)
Lymphoedema (Vascular disorders) | 4/36 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days